CLINICAL TRIAL: NCT00626015
Title: Zenapax®-Activated Peptide ImmunoTherapy [ZAP IT]
Brief Title: Chemotherapy, Radiation Therapy, and Vaccine Therapy With Basiliximab in Treating Patients With Glioblastoma Multiforme That Has Been Removed by Surgery
Acronym: ZAP IT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Sampson (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, John Sampson, Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000947; R21CA132891 (NIH); CDR0000579573 (Other: National Cancer Institute)
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Malignant Neoplasms of Brain
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult high grade glioma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Glioma | interventions — Daclizumab; Temozolomide; rindopepimut

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (Experimental): Temozolomide, PEP-3-KLH conjugate vaccine, and daclizumab
  Interventions: Biological: PEP-3-KLH conjugate vaccine; Biological: daclizumab; Drug: temozolomide
- Arm II (Experimental): Temozolomide, PEP-3-KLH conjugate vaccine, and normal saline
  Interventions: Biological: PEP-3-KLH conjugate vaccine; Drug: temozolomide; Other: placebo
- Basiliximab (Experimental): Patients will receive basiliximab 20 mg IV with vaccine # 1 only and continue with PEP-3-KLH, temozolomide.
  Interventions: Biological: PEP-3-KLH

INTERVENTIONS:
Biological: PEP-3-KLH conjugate vaccine — Given intradermally
  Arms: Arm I; Arm II
Biological: daclizumab — Given IV
  Arms: Arm I
Drug: temozolomide — Given by mouth.
  Arms: Arm I; Arm II
Other: placebo — Given IV
  Arms: Arm II
Biological: PEP-3-KLH — Basiliximab 20 mg IV over 30 minutes with PEP-3-KLH vaccine # 1 only.
  Other Names: CDX-110; EGFRvIII-KLH
  Arms: Basiliximab

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Vaccines may help the body build an effective immune response to kill tumor cells. Monoclonal antibodies, such as basiliximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving chemotherapy, radiation therapy, and vaccine therapy together with basiliximab is a more effective treatment for glioblastoma multiforme than chemotherapy, radiation therapy, and vaccine therapy alone.

PURPOSE: This randomized phase I trial is studying the side effects and best way to give chemotherapy and radiation therapy followed by vaccine therapy with basiliximab in treating patients with glioblastoma multiforme that has been removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if basiliximab inhibits the functional and numeric recovery of T-regulatory cells (Tregs) after therapeutic temozolomide (TMZ)-induced lymphopenia in the context of vaccinating adult patients with newly diagnosed glioblastoma multiforme (GBM) using PEPvIII-keyhole limpet hemocyanin (KLH).

Secondary

* To evaluate the safety of basiliximab in the context of vaccinating adult patients with newly diagnosed GBM using PEP-3-KLH conjugate vaccine during recovery from therapeutic TMZ-induced lymphopenia.
* To determine if basiliximab enhances the magnitude or character of PEPvIII-KLH-induced cellular or humoral immune responses, inhibits or enhances activation-induced cell death, or induces immunologic or clinical evidence of autoimmunity.
* To determine if basiliximab enhances the magnitude or character of PEPvIII-KLH-induced cellular or humoral immune responses, inhibits or enhances activation-induced cell death, or induces immunologic or clinical evidence of autoimmunity.
* To determine if basiliximab alters the phenotype (CD56-expression), cytokine secretion profile, or cytotoxicity of CD3-negative CD56-positive natural killer cells.
* To determine if basiliximab, in addition to vaccination, extend progression-free survival compared to historical cohorts.
* To characterize immunologic cell infiltrate in recurrent tumors and seek evidence of antigen escape outgrowth.

OUTLINE:

* Leukapheresis: Patients undergo leukapheresis over 2-4 hours for immunologic monitoring.
* Concurrent standard adjuvant chemoradiotherapy: Patients receive external-beam radiotherapy once daily, 5 days a week, over 6-7 weeks (33 fractions) and concurrent temozolomide by mouth 7 days a week for up to 49 days beginning on the first day and continuing until the last day of radiotherapy.
* Temozolomide and PEP-3-KLH conjugate vaccine: Approximately 3 weeks after completion of radiotherapy, patients receive temozolomide by mouth on days 1-21, or on days 1-5 depending on their treating neuro-oncologist, basiliximab IV over 30 minutes on day 21, and PEP-3-KLH conjugate vaccine intradermally on days 21, 35, and 49.

Patients then receive a second course of temozolomide by mouth on days 1-21 or days 1-5, depending on their treating neuro-oncologist. Treatment with temozolomide repeats every 4 weeks for 5 additional courses. Patients also receive PEP-3-KLH conjugate vaccine on day 21 of each remaining temozolomide course. Patients then receive the vaccine monthly until disease progression.

Patients undergo blood sample collection periodically for laboratory studies.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histopathologic diagnosis of WHO grade III or WHO grade IV high grade glioma

  * Newly diagnosed disease
* Meets the following criteria:

  * The patient must undergo leukapheresis for immunologic monitoring
* Tumor expression of EGFRvIII by immunohistochemistry (IHC) or polymerase chain reaction (PCR)
* No radiographic or cytologic evidence of leptomeningeal or multicentric disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status ≥ 80%
* Curran Group status of I-IV
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No conditions that will potentially confound the study results, including any of the following:

  * Active infection requiring treatment or an unexplained febrile (> 101.5°F) illness
  * Known immunosuppressive disease or known HIV infection
  * Unstable or severe intercurrent medical conditions such as severe heart or lung disease
* No demonstrated allergy to TMZ
* Able to tolerate TMZ

  * TMZ-induced lymphopenia allowed
* No prior allergic reaction to daclizumab/basiliximab or its components

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other conventional therapeutic intervention other than steroids, radiation, or temozolomide (TMZ) prior to enrollment
* No prior allogeneic solid organ transplantation
* No prior inguinal lymph node dissection, radiosurgery, brachytherapy, or radiolabeled monoclonal antibodies
* No corticosteroids at a dose above physiologic level except nasal or inhaled steroid at the time of first study vaccination

  * For the purposes of this study, physiologic dose is defined as < 2 mg of dexamethasone/day
  * Once study vaccinations have been initiated, if patients subsequently require increased steroids, they are permitted to remain on the study
* No prior daclizumab/basiliximab

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Functional suppressive capacity of CD4+CD25+CD127- T-regulatory cells | 26 months
Comparison of proliferative T-cell response to phytohemagglutinin (PHA) among treatment groups (with versus without daclizumab/basiliximab) | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Duane Mitchell, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Sampson JH, Schmittling RJ, Archer GE, Congdon KL, Nair SK, Reap EA, Desjardins A, Friedman AH, Friedman HS, Herndon JE 2nd, Coan A, McLendon RE, Reardon DA, Vredenburgh JJ, Bigner DD, Mitchell DA. A pilot study of IL-2Ralpha blockade during lymphopenia depletes regulatory T-cells and correlates with enhanced immunity in patients with glioblastoma. PLoS One. 2012;7(2):e31046. doi: 10.1371/journal.pone.0031046. Epub 2012 Feb 27. PMID 22383993